CLINICAL TRIAL: NCT06717581
Title: Variation in Drug Interactions in People With HIV (PLWH) Aged 60 Years and Older on Stable Antiretroviral Therapy Making a Switch to Bictegravir/Tenofovir Alafenamide/Emtricitabine
Brief Title: Variation in Drug Interactions in People With HIV (PLWH) Aged 60 Years and Older.
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: BICTER
Record Dates: First submitted 2024-12-01; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: HIV Infections; Drug Interaction; Elderly Infection; Comorbidities and Coexisting Conditions; Cardiovascular Diseases; Metabolic Disease; Renal Disease; Osteoporosis Risk; Neoplasms
Keywords: HIV; Drug Interactions; Retrovirus; Comorbidities
MeSH Terms: conditions — HIV Infections; Cardiovascular Diseases; Metabolic Diseases; Kidney Diseases; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | US Export: No

GROUPS / COHORTS (1):
- people with HIV (PLWH) aged 60 years and older: people with HIV (PLWH) aged 60 years and older on stable antiretroviral therapy who switch to bictegravir/tenofovir alafenamide/emtricitabine.

SUMMARY:
Several cohort studies have recently shown a significant increase in the mean age of PLWH ( People Living With HIV) and in the prevalence of people in advanced age in the various cohorts, as a result of the marked increase in the mean life expectancy of these people achieved by modern antiretroviral combination therapies.

However, the high prevalence of comorbidities exposes PLWH in old age to the need to take multiple drug treatments in addition to antiretroviral therapy, with the gradually increasing risk of unfavorable pharmacokinetic interactions between antiretroviral drugs and drugs taken to treat the comorbidities.

This project consists of an observational, cohort, retrospective, single-center study and aims to evaluate the variation in the number and type of clinically significant drug interactions between antiretroviral therapy and concomitant therapies in PLWH aged >60 years on stable antiretroviral therapy who, for any reason at the Clinician's discretion, have made a switch from ongoing antiretroviral therapy to the bictegravir/emtricitabine/tenofovir alafenamide regimen.

DETAILED DESCRIPTION:
The introduction of integrase inhibitors into clinical practice has greatly improved the efficacy and tolerability of modern antiretroviral combination therapies for the treatment of patients with HIV-1 infection. Indeed, these drugs have shown in registration studies high antiviral potency associated with a negligible incidence of short- and long-term adverse events, so much so that they are consistently included in the drug regimens recommended by all international guidelines for the treatment of HIV-positive patients naive to antiretroviral therapy.

Several cohort studies have recently shown a significant increase in the mean age of PLWH ( People Living With HIV) and in the prevalence of people in advanced age in the various cohorts, as a result of the marked increase in the mean life expectancy of these people achieved by modern antiretroviral combination therapies.

PLWH in advanced age, however, have a high prevalence of noninfectious comorbidities (cardiovascular disease, metabolic abnormalities, chronic renal failure, osteopenia-osteoporosis, neoplastic diseases, etc.), brought about by age-related aging but also by their accelerated biological aging caused by HIV infection and associated chronic inflammation and immunoactivation.

The high prevalence of comorbidities exposes PLWH in old age to the need to take multiple drug treatments in addition to antiretroviral therapy, with the gradually increasing risk of unfavorable pharmacokinetic interactions between antiretroviral drugs and drugs taken to treat the comorbidities.

The effect of such interactions can be either a reduction in plasma concentrations with reduced efficacy of antiretroviral drugs or an increase in plasma levels of concomitant drugs and the risk of toxicity induced by them.

The availability of integrase inbitors such as bictegravir, i.e., antiretroviral drugs characterized by a very low risk of drug interactions (because they are generally not metabolized by hepatic cytochrome P450 3A4 isoenzymes), has made it possible to significantly reduce the risk of interactions between antiretroviral therapy and concomitant therapy, especially in people of advanced age, while providing high viro-immunologic efficacy and a favorable effect on the cardio-metabolic profile.

This project consists of an observational, cohort, retrospective, single-center study and aims to evaluate the variation in the number and type of clinically significant drug interactions between antiretroviral therapy and concomitant therapies in PLWH aged >60 years on stable antiretroviral therapy who, for any reason at the Clinician's discretion, have made a switch from ongoing antiretroviral therapy to the bictegravir/emtricitabine/tenofovir alafenamide regimen.

ELIGIBILITY:
Inclusion Criteria:

* Age > 60 years
* Non-infectious comorbidities receiving drug therapy
* Receiving BIC/TAF/FTC therapy at the time of of enrollment

Exclusion Criteria:

* Genotypic resistance testing that present or past evidence of viral resistance to the integrase inhibitor class, to emtricitabine or to tenofovir
* Severe acute infectious disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study involves the enrollment of 50 patients (number calculated on the basis of the patient's medical history with the main characteristics for the purpose of enrollment in the clinical trial) who will be seen at the outpatient clinics of the Infectious Diseases Operative Unit of the IRCCS, Azienda Ospedaliero Universitaria di Bologna Policlinico di Sant'Orsola, during the period from January 1, 2021 to December 31, 2022.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2025-04-11 (Estimated); Study Completion 2025-10-11 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the change in the total number of clinically significant drug-drug interactions (DDIs) | 12 Months
  Evaluation of the change in the total number of clinically significant drug-drug interactions (DDIs) between antiretroviral drugs and concomitant drugs following therapeutic switch to bictegravir/emtricitabine/tenofovir alafenamide.
Evaluation of the change in the number of clinically significant DDIs between antiretroviral drugs and drugs of specific therapeutic classes | 12 Months
  Evaluation of the change in the number of clinically significant DDIs between antiretroviral drugs and drugs of specific therapeutic classes (cardiovascular, hypolipidemic, hypoglycemic, neurological/psychiatric, etc.) following therapeutic switch to bictegravir/emtricitabine/tenofovir alafenamide

SECONDARY OUTCOMES:
Evaluation of viro-immunological parameters and incidence of clinical adverse events and treatment discontinuations | 12 Months
  Evaluation of viro-immunological parameters and incidence of clinical adverse events and treatment discontinuations during the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Calza, Medicine, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Yes
The investigator agrees to make the results public at the end of the study. For this purpose, the study will be registered on an Open Science platform. Any formal submission or publication of data derived from this study should be understood as a publication by the Investigator.
Supporting Information: SAP, CSR, Analytic Code
Time Frame: 12 Months
Access Criteria: Any formal submission or publication of data derived from this study should be understood as a publication by the Investigator.

REFERENCES:
- [Background] McIntosh RC, Ironson G, Antoni M, Kumar M, Fletcher MA, Schneiderman N. Alexithymia is linked to neurocognitive, psychological, neuroendocrine, and immune dysfunction in persons living with HIV. Brain Behav Immun. 2014 Feb;36:165-75. doi: 10.1016/j.bbi.2013.10.024. Epub 2013 Nov 1. PMID 24184475
- [Background] Pompili M, Pennica A, Serafini G, Battuello M, Innamorati M, Teti E, Girardi N, Amore M, Lamis DA, Aceti A, Girardi P. Depression and affective temperaments are associated with poor health-related quality of life in patients with HIV infection. J Psychiatr Pract. 2013 Mar;19(2):109-17. doi: 10.1097/01.pra.0000428557.56211.cf. PMID 23507812
- [Background] Parruti G, Vadini F, Sozio F, Mazzott E, Ursini T, Polill E, Di Stefano P, Tontodonati M, Verrocchio MC, Fulcheri M, Calella G, Santilli F, Manzoli L. Psychological factors, including alexithymia, in the prediction of cardiovascular risk in HIV infected patients: results of a cohort study. PLoS One. 2013;8(1):e54555. doi: 10.1371/journal.pone.0054555. Epub 2013 Jan 22. PMID 23349927
- [Background] Leyro TM, Vujanovic AA, Bonn-Miller MO. Examining associations between cognitive-affective vulnerability and HIV symptom severity, perceived barriers to treatment adherence, and viral load among HIV-positive adults. Int J Behav Med. 2015 Feb;22(1):139-48. doi: 10.1007/s12529-014-9404-8. PMID 24643444
- [Background] McIntosh RC, Ironson G, Antoni M, Fletcher MA, Schneiderman N. Alexithymia, Assertiveness and Psychosocial Functioning in HIV: Implications for Medication Adherence and Disease Severity. AIDS Behav. 2016 Feb;20(2):325-38. doi: 10.1007/s10461-015-1126-7. PMID 26143246